CLINICAL TRIAL: NCT01856751
Title: Use of a TGA and TEM in the Assessment of the Efficacy of Treatment With APCC or rFVIIa Concentrate in Patients With Acquired Haemophilia and in Patients With Haemophilia A With Inhibitors
Brief Title: Use of a TGA and TEM in the Assessment of the Efficacy of Treatment With APCC or rFVIIa
Acronym: Thrombus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stowarzyszenie Pomocy Chorym na Zakrzepicę i Skazy Krwotoczne Thrombus (Other)
Responsible Party: Sponsor
Other Study IDs: TGA-TEM
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Haemophilia
Keywords: Haemophilia; TGA; TEM
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — this data is not applicable
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- haemophilia: Patients with acquired haemophilia. Patients with haemophilia A with inhibitor.

SUMMARY:
Occurrence of inhibitors to coagulation factor VIII is diagnosed in ~30% patients with haemophilia A. Presence of inhibitor with a titre >5 BU/ml requires the use of by-passing agents: recombinant activated Factor VIIa concentrate (rFVIIa) and/or activated prothrombin complex concentrate (APCC). Similarly, haemorrhagic complications in patients with acquired haemophilia and inhibitor titre >5 BU/ml should be treated with by-passing agents.

Response to treatment with by-passing agents is patient-specific, and can vary in the same patient during subsequent bleedings. Some patients have good response to both products, however in other patients a better bleeding control is provided by one of the mentioned above agents (APCC or rFVIIa). There are clinical situations when severe bleedings requires an alternate use of both these agents.

Traditional methods of laboratory tests used post-treatment in patients with haemophilia without inhibitors are useless in the presence of inhibitor. Laboratory monitoring of therapy with by-passing agents is possible with the use of global tests for the coagulation process assessment, which are as follows: thrombin generation assay (TGA) and thromboelastometry (TEM).

Several studies revealed that TGA allows a monitoring of therapy with by-passing agents in patients with haemophilia A and inhibitor - the choice of the most effective treatment option - agent type and its dose, as well as laboratory assessment of treatment efficacy.

Up to date, laboratory tests assessing the efficacy of by-passing agents in patients with acquired haemophilia were not conducted.

In Factor VIII or IX deficiency conditions, fibrin's fibres generated by thrombin are morphologically thicker, and blood clots have increased susceptibility to fibrinolytic enzymes. Blood clot stability may be assessed with the use of thromboelastometry (TEM). We can hypothesize that simultaneous use of TGA and TEM methods may allow for an assessment of patient's individual response to therapy with by-passing agents. Clinical significance of the minimal dose of APCC and rFVIIa, needed to TGA and TEM normalization, requires further studies.

Tests' purpose: Examination of the hypothesis that simultaneous use of thrombin generation assay (TGA) and thromboelastometry (TEM) may facilitate the choice of optimal therapy with by-passing agents and laboratory monitoring of efficacy of those agents in patients with acquired haemophilia or haemophilia A with inhibitor.

DETAILED DESCRIPTION:
This section is Not applicable

ELIGIBILITY:
Inclusion Criteria:

* patients with acquired haemophilia
* patients with congenital haemophilia A with inhibitor

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with acquired haemophilia 20 patients with congenital haemophilia A with inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of patient's individual response to therapy with by-passing agents by simultaneous use of TGA and TEM methods. | 48 hours
  This is non-inverventional study as the protocol will not assign specific treatment to the particular subjects of the study. Patients will be treated with APCC or rFVIIa based on the experience of the study site. Patients are prescribed a treatment according to their physician's judgement or local clinical practice. This is observation of the everyday clinical practise on site.

CONTACTS AND LOCATIONS:
Overall Officials: Krystyna Zawilska, MD, PhD, Principal Investigator — Centrum Diagnostyczno - Lecznicze INTERLAB; Maria Podolak-Dawidziak, MD,PhD, Principal Investigator — Katedra i Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Akademia Medyczna; Andrzej Mital, MD, PhD, Principal Investigator — Katedra i Klinika Hematologii i Transplantologii Gdanski Uniwersytet Medyczny; Jerzy Windyga, MD, PhD, Principal Investigator — Instytut Hematologii i Transfuzjologii w Warszawie; Krzysztof Chojnowski, MD, PhD, Principal Investigator — Klinika Hematologii Uniwersytetu Medycznego w Lodzi Wojewodzki Szpital Specjalistyczny im. M. Kopernika; Jacek Musial, MD, PhD, Principal Investigator — Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Alergii i Immunologii
Locations (6):
- Poland (6):
  - Katedra i Klinika Hematologii i Transplantologii Gdanski Uniwersytet Medyczny, Gdansk
  - Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Alergii i Immunologii, Krakow
  - Klinika Hematologii Uniwersytetu Medycznego w Lodzi Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Centrum Diagnostyczno - Lecznicze INTERLAB, Poznan
  - Instytut Hematologii i Transfuzjologii w Warszawie, Warsaw
  - Katedra i Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Akademia Medyczna, Wroclaw

REFERENCES:
- [Background] Dargaud Y, Negrier C. Thrombin generation testing in haemophilia comprehensive care centres. Haemophilia. 2010 Mar;16(2):223-30. doi: 10.1111/j.1365-2516.2009.02082.x. Epub 2009 Aug 27. PMID 19719549
- [Background] Berntorp E. Differential response to bypassing agents complicates treatment in patients with haemophilia and inhibitors. Haemophilia. 2009 Jan;15(1):3-10. doi: 10.1111/j.1365-2516.2008.01931.x. Epub 2008 Nov 10. PMID 19016901
- [Background] Dargaud Y, Bordet JC, Lienhart A, Negrier C. Use of the thrombin generation test to evaluate response to treatment with recombinant activated factor VII. Semin Hematol. 2008 Apr;45(2 Suppl 1):S72-3. doi: 10.1053/j.seminhematol.2008.03.008. No abstract available. PMID 18544431
- [Background] Livnat T, Martinowitz U, Zivelin A, Seligsohn U. Effects of factor VIII inhibitor bypassing activity (FEIBA), recombinant factor VIIa or both on thrombin generation in normal and haemophilia A plasma. Haemophilia. 2008 Jul;14(4):782-6. doi: 10.1111/j.1365-2516.2008.01688.x. Epub 2008 Mar 21. PMID 18371162